CLINICAL TRIAL: NCT06303128
Title: Penicillin Allergy Delabeling After a One-Dose Versus Two-Dose Graded Direct Oral Challenge
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: James Tarbox, MD (Other)
Collaborators: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor-Investigator, James Tarbox, MD, Associate Professor, Texas Tech University Health Sciences Center
Organization: Texas Tech University Health Sciences Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: IRB-FY2024-61
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Penicillin Allergy
Keywords: low-risk allergy; amoxicillin; drug allergy; direct oral challenge
MeSH Terms: conditions — Drug Hypersensitivity | interventions — Amoxicillin; Population Groups; WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Intervention Model Description: - Low-risk penicillin allergic patients ("low-risk" determined by a PEN-FAST score of 2 or less) will be recruited. Clinically stable patients will be randomly assigned in a double-blinded manner to receive either a one-dose or graded two-dose direct oral challenge with amoxicillin in an outpatient setting. Those assigned to receive one dose of amoxicillin will receive a placebo in place of a second dose of amoxicillin. Both groups will receive the same cumulative dose of amoxicillin (250mg) by the end of the trial. Baseline vital signs will be obtained and tracked throughout the trial. Patients will also be monitored for development of signs of allergic reactions during the trial, with administration of appropriate treatment should the need arise.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- One-dose group (Experimental): Patients assigned to this group will receive a liquid placebo followed by full-dose liquid amoxicillin 250mg PO thirty minutes later.
  Interventions: Drug: Amoxicillin 250 MG; Drug: Placebo
- Graded, two-dose group (Active Comparator): Patients assigned to this group will receive liquid amoxicillin (25% of 250mg dose), followed by liquid amoxicillin 187.5mg PO (75% of 250mg dose) thirty minutes later.
  Interventions: Drug: Amoxicillin 62.5mg; Drug: Amoxicillin 187.5mg

INTERVENTIONS:
Drug: Amoxicillin 250 MG — Liquid amoxicillin 250mg PO
  Other Names: One-dose group
  Arms: One-dose group
Drug: Placebo — Given prior to amoxicillin 250mg in one-dose group
  Other Names: Liquid placebo (Syrpalta or similar) for one-dose group
  Arms: One-dose group
Drug: Amoxicillin 62.5mg — Given first in two-dose group, liquid amoxicillin 62.5mg PO
  Other Names: Two-dose group, dose 1 of 2
  Arms: Graded, two-dose group
Drug: Amoxicillin 187.5mg — Given second in two-dose group, liquid amoxicillin 187.5mg PO
  Other Names: Two-dose group, dose 2 of 2
  Arms: Graded, two-dose group

SUMMARY:
The goal of this clinical trial is to learn about dosing when testing to see if a penicillin allergy label can be removed from adults that had been labeled as "penicillin-allergic" previously. The main question it aims to answer is:

- In penicillin-allergic patients that are at low risk of having an allergic reaction, is a one-dose oral challenge with amoxicillin (a penicillin-based antibiotic) as safe and effective as a two-dose oral challenge?

Participants will, after being identified as having a low-risk penicillin allergy, be administered oral amoxicillin in a controlled setting and then monitored for an allergic reaction. Researchers will compare participants that took one dose of amoxicillin to participants that took two doses of amoxicillin (a small dose and then a larger dose) to see if either group was more likely to develop an allergic reaction.

DETAILED DESCRIPTION:
Anywhere from 5-15% of patients have a reported penicillin allergy listed in their medical record. However, most patients with this listed allergy had reactions with characteristics that would qualify their penicillin allergy as low-risk of having a subsequent serious reaction (when considering initial reaction symptoms, time since initial reaction and if treatment was required). Of patients with penicillin allergy listed, it has been demonstrated that >90% can tolerate penicillin after further evaluation, indicating a significant number of patients with an unnecessary penicillin allergy label.

Penicillin allergy delabeling is a practice commonly performed by allergists to test patients for safe removal of penicillin allergy from their medical records. The protocol of penicillin allergy delabeling has historically consisted of a skin test, followed by a two-step graded direct oral challenge, in which patients are given a smaller, then larger, oral dose of amoxicillin, a penicillin-containing medication. The patient is monitored closely throughout the process for reaction to penicillin and, if necessary, treatment is given for management of reaction symptoms. This method, though functional, takes time and resources to delabel patients.

As our understanding of penicillin drug allergy evolves, it may be possible to reduce the number of steps (and therefore resources) necessary to safely remove penicillin allergy labels. New data suggests that skin testing may not be a necessary step in penicillin allergy delabeling in a subset of low-risk patients. It has also been demonstrated in several studies that a single-dose direct oral challenge (rather than a two-step graded dose) is safe. A recent pilot study also showed that penicillin allergy delabeling can be safely performed in a primary care setting without the direct supervision of an allergist.

Per the authors' literature review, no prospective studies have directly compared the safety and efficacy of a single-dose versus a two-dose graded direct oral challenge. We propose a non-inferiority study in which patients classified as having a low-risk penicillin allergy are randomized into two groups and then receive either a single-dose or the traditional two-dose graded direct oral challenge to be able to evaluate these two treatment protocols in a side-by-side fashion. The results will contribute to our understanding of if a single-dose direct oral challenge can be safely used in place of the traditional two-dose graded direct oral challenge, thus reducing barriers for implementation in a primary care setting.

Patients with penicillin allergy that express interest through publicly posted recruitment materials will be screened to determine if they meet criteria for a "low-risk" allergy through the PEN-FAST screening tool, a recently developed, externally validated penicillin allergy risk assessment calculator. Those that meet the low-risk criteria and other eligibility criteria will be scheduled for an outpatient delabeling appointment. Participants will be randomly assigned in a double-blinded manner to receive either a two-dose graded direct oral challenge (DOC) with amoxicillin or a one-dose DOC placebo, followed by amoxicillin. Each group will receive the same cumulative dose of amoxicillin by the end of the challenge. Participants assigned to the two-dose graded DOC will be administered 62.5mg amoxicillin (25% of the full dose), followed by 187.5mg amoxicillin. Patients assigned to the one-dose DOC will be administered a placebo (Syrpalta or similar, a syrup used in drug compounding), followed by 250mg amoxicillin.

Doses will be given 30 minutes apart from one another. Both groups will be observed for a minimum of 1 hour after administration of the final dose of amoxicillin. Vital signs will be taken immediately before starting the trial, 30 minutes after administration of the first dose, and 60 minutes after administration of the second dose. If patients develop a reaction at any point in the trial, they will be treated according to the type and severity of their symptoms in an appropriate and standardized manner.

As both single-dose and graded two-dose challenges have been used in clinical practice to remove penicillin allergy labels in the past, if no reaction occurs, patients can have their penicillin allergy removed from their chart. Patients will be contacted around 5 days after the challenge to evaluate for any delayed reactions. If, at the 5-day phone call, patients have not had any other reactions suspected to be related to amoxicillin, their penicillin allergy label will be removed at that time. Patients will also be contacted around 6 months after the DOC to evaluate for any reactions to antibiotics received since successful delabeling. The two groups will then be compared to determine if the one-dose challenge is noninferior to the standard graded two-dose challenge (based upon the rate of successful delabeling without adverse reactions).

Currently, this study is approved as a single-site study only.

ELIGIBILITY:
Inclusion Criteria:

* Expresses interest in participating by calling or filling out information form on study website
* Reports an allergy to one of the following medications: penicillin VK, penicillin G, amoxicillin, ampicillin, dicloxacillin, flucloxacillin, nafcillin, oxacillin, amoxicillin- clavulanate, ampicillin-sulbactam. Subjects with an unspecified penicillin allergy are also eligible to participate.

Exclusion Criteria:

* Penicillin allergy deemed to be more than "low-risk" per PEN-FAST (score ≥ 3 points)
* History of acute kidney injury (acute interstitial nephritis), severe liver impairment (drug- induced liver injury), serum sickness, or isolated drug fever attributed to a penicillin- based antibiotic
* Anaphylaxis for any reason in the last year
* Cognitive impairment where a collateral history could not be obtained and/or patient does not have capacity to consent for themselves
* Pregnant (self-reported)
* Any illness or condition that would increase the risk of participation in the study, per the evaluating clinician's judgment
* Active treatment of or history of acute angle closure glaucoma
* On H1- or H2-blockers (i.e. diphenhydramine, hydroxyzine, chlorpheniramine, cetirizine, levocetirizine, loratadine, fexofenadine or famotidine, ranitidine, cimetidine, nizatidine, respectively) within 72 hours of initiating direct oral challenge (will be counseled to discontinue prior to testing)
* Actively receiving greater than stress dose steroid (hydrocortisone >50mg four times a day or steroid equivalent)
* Actively receiving any antibiotic
* Relative contraindication: Patients on beta blockers and angiotensin converting enzyme inhibitors (ACE inhibitors) will have an open dialog with the study team regarding the risks and benefits of testing a low-risk penicillin allergy patient. A joint decision will be made based on the patient's preference and the physician's comfort level.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2024-02-03 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of successfully "delabeled" subjects in one-dose versus two-dose groups | 5 days (at time of first follow up phone call)
  Percentage of subjects that successfully complete either the one-dose or graded two-dose direct oral challenge with amoxicillin without adverse reactions during the challenge, as determined by no reaction reported at first follow up phone call.

SECONDARY OUTCOMES:
Analysis of adverse reactions | 2 hours (during direct oral challenge) and 5 days (at time of first follow up phone call)
  Percentage of subjects that report adverse reactions during direct oral challenge and at 5-day follow-up phone call, including type of reaction, timing, severity, treatment required (if any), and classification of degree of causality.
Analysis of medical and allergic history | Reported at time of direct oral challenge
  For further stratification of primary outcome, other medical and allergic history items including: reported penicillin allergy label, history of cephalosporin allergy, PEN-FAST score, time (in years) since index reaction, time (in hours) between administration of medication and index reaction, treatment required for index reaction, antibiotics tolerated since index reaction, history of other atopic conditions, and use of beta blockers/ACE inhibitors.
Validation of penicillin allergy delabeling | 6 months
  Data from 6-month follow up phone call including: percentage of successfully delabeled patients able to tolerate penicillin-derived antibiotics since DOC and any associated reactions, percentage of patients confident in taking a penicillin derivative should it be required in the future.
Analysis of demographic data | Reported at time of direct oral challenge
  For further stratification of primary outcome, demographic data, including age, gender, race/ethnicity, urban vs. rural and other measures of socioeconomic status. This will allow us to analyze differences in reaction rates between different groups, as well as psychological differences between groups when considering patient confidence in their allergy label being removed.

CONTACTS AND LOCATIONS:
Overall Officials: James A Tarbox, MD, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article that is planned to be published, after deidentification.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal to achieve aims in the approved proposal.

REFERENCES:
- [Background] Blumenthal KG, Peter JG, Trubiano JA, Phillips EJ. Antibiotic allergy. Lancet. 2019 Jan 12;393(10167):183-198. doi: 10.1016/S0140-6736(18)32218-9. Epub 2018 Dec 14. PMID 30558872
- [Background] Trubiano JA, Vogrin S, Chua KYL, Bourke J, Yun J, Douglas A, Stone CA, Yu R, Groenendijk L, Holmes NE, Phillips EJ. Development and Validation of a Penicillin Allergy Clinical Decision Rule. JAMA Intern Med. 2020 May 1;180(5):745-752. doi: 10.1001/jamainternmed.2020.0403. PMID 32176248
- [Background] Khan DA, Banerji A, Blumenthal KG, Phillips EJ, Solensky R, White AA, Bernstein JA, Chu DK, Ellis AK, Golden DBK, Greenhawt MJ, Horner CC, Ledford D, Lieberman JA, Oppenheimer J, Rank MA, Shaker MS, Stukus DR, Wallace D, Wang J; Chief Editor(s):; Khan DA, Golden DBK, Shaker M, Stukus DR; Workgroup Contributors:; Khan DA, Banerji A, Blumenthal KG, Phillips EJ, Solensky R, White AA; Joint Task Force on Practice Parameters Reviewers:; Bernstein JA, Chu DK, Ellis AK, Golden DBK, Greenhawt MJ, Horner CC, Ledford D, Lieberman JA, Oppenheimer J, Rank MA, Shaker MS, Stukus DR, Wallace D, Wang J. Drug allergy: A 2022 practice parameter update. J Allergy Clin Immunol. 2022 Dec;150(6):1333-1393. doi: 10.1016/j.jaci.2022.08.028. Epub 2022 Sep 17. No abstract available. PMID 36122788
- [Background] Iammatteo M, Lezmi G, Confino-Cohen R, Tucker M, Ben-Shoshan M, Caubet JC. Direct Challenges for the Evaluation of Beta-Lactam Allergy: Evidence and Conditions for Not Performing Skin Testing. J Allergy Clin Immunol Pract. 2021 Aug;9(8):2947-2956. doi: 10.1016/j.jaip.2021.04.073. PMID 34366093
- [Background] Iammatteo M, Alvarez Arango S, Ferastraoaru D, Akbar N, Lee AY, Cohen HW, Jerschow E. Safety and Outcomes of Oral Graded Challenges to Amoxicillin without Prior Skin Testing. J Allergy Clin Immunol Pract. 2019 Jan;7(1):236-243. doi: 10.1016/j.jaip.2018.05.008. Epub 2018 May 23. PMID 29802906
- [Background] Copaescu AM, Vogrin S, James F, Chua KYL, Rose MT, De Luca J, Waldron J, Awad A, Godsell J, Mitri E, Lambros B, Douglas A, Youcef Khoudja R, Isabwe GAC, Genest G, Fein M, Radojicic C, Collier A, Lugar P, Stone C, Ben-Shoshan M, Turner NA, Holmes NE, Phillips EJ, Trubiano JA. Efficacy of a Clinical Decision Rule to Enable Direct Oral Challenge in Patients With Low-Risk Penicillin Allergy: The PALACE Randomized Clinical Trial. JAMA Intern Med. 2023 Sep 1;183(9):944-952. doi: 10.1001/jamainternmed.2023.2986. PMID 37459086
- [Background] Wang LA, Patel K, Kuruvilla ME, Shih J. Direct amoxicillin challenge without preliminary skin testing for pediatric patients with penicillin allergy labels. Ann Allergy Asthma Immunol. 2020 Aug;125(2):226-228. doi: 10.1016/j.anai.2020.05.004. Epub 2020 May 11. No abstract available. PMID 32407949
- [Background] Lin L, Nagtegaal JE, Buijtels PCAM, Jong E. Antimicrobial stewardship intervention: optimizing antibiotic treatment in hospitalized patients with reported antibiotic allergy. J Hosp Infect. 2020 Feb;104(2):137-143. doi: 10.1016/j.jhin.2019.10.007. Epub 2019 Oct 13. PMID 31618608
- [Background] Trubiano JA, Smibert O, Douglas A, Devchand M, Lambros B, Holmes NE, Chua KY, Phillips EJ, Slavin MA. The Safety and Efficacy of an Oral Penicillin Challenge Program in Cancer Patients: A Multicenter Pilot Study. Open Forum Infect Dis. 2018 Nov 17;5(12):ofy306. doi: 10.1093/ofid/ofy306. eCollection 2018 Dec. PMID 30547046
- [Background] Chua KYL, Vogrin S, Bury S, Douglas A, Holmes NE, Tan N, Brusco NK, Hall R, Lambros B, Lean J, Stevenson W, Devchand M, Garrett K, Thursky K, Grayson ML, Slavin MA, Phillips EJ, Trubiano JA. The Penicillin Allergy Delabeling Program: A Multicenter Whole-of-Hospital Health Services Intervention and Comparative Effectiveness Study. Clin Infect Dis. 2021 Aug 2;73(3):487-496. doi: 10.1093/cid/ciaa653. PMID 32756983
- [Background] Tucker MH, Lomas CM, Ramchandar N, Waldram JD. Amoxicillin challenge without penicillin skin testing in evaluation of penicillin allergy in a cohort of Marine recruits. J Allergy Clin Immunol Pract. 2017 May-Jun;5(3):813-815. doi: 10.1016/j.jaip.2017.01.023. Epub 2017 Mar 21. No abstract available. PMID 28341170
- [Background] Kuruvilla M, Shih J, Patel K, Scanlon N. Direct oral amoxicillin challenge without preliminary skin testing in adult patients with allergy and at low risk with reported penicillin allergy. Allergy Asthma Proc. 2019 Jan 1;40(1):57-61. doi: 10.2500/aap.2019.40.4184. PMID 30582497
- [Background] Chow TG, Patel G, Mohammed M, Johnson D, Khan DA. Delabeling penicillin allergy in a pediatric primary care clinic. Ann Allergy Asthma Immunol. 2023 May;130(5):667-669. doi: 10.1016/j.anai.2023.01.034. Epub 2023 Feb 2. No abstract available. PMID 36738783
- [Background] Livirya S, Pithie A, Chua I, Hamilton N, Doogue M, Isenman H. Oral amoxicillin challenge for low-risk penicillin allergic patients. Intern Med J. 2022 Feb;52(2):295-300. doi: 10.1111/imj.14978. Epub 2022 Jan 12. PMID 32672891
- See also: Recruiting Website — https://delabelingpenicillin.wixsite.com/penicillin-de-labeli